CLINICAL TRIAL: NCT05113173
Title: Study on the Relationship Between Different Pathological Features of Achalasia and Prognosis of Per-oral Endoscopic Myotomy
Brief Title: Study on the Relationship Between Pathological Features of Achalasia and Prognosis of Per-oral Endoscopic Myotomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fandong Meng (Other)
Responsible Party: Sponsor-Investigator, Fandong Meng, chief physician, Beijing Friendship Hospital
Organization: Beijing Friendship Hospital (Other)
Other Study IDs: YYYXYJ-2021-085
Record Dates: First submitted 2021-10-11; First posted 2021-11-09 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Achalasia
Keywords: Esophageal Achalasia; per-oral endoscopic myotomy; pathology
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — esophageal muscular layers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type I Achalasia: Severe loss of ganglion cells,loss of ICCs.
- Type II Achalasia: Loss of ICCs, mild loss of ganglion cells.
- Type III Achalasia: Preserved ICCs, less loss of ganglion.

SUMMARY:
Achalasia is the most common motility disorder of esophagus, characterized by disorders of the lower esophageal sphincter (LES). Normal peristalsis of the esophagus is eliminated and replaced by synchronous or ineffective contraction. Based on high-resolution manometry (HRM), the participants with achalasia were categorized into 3 subtypes, type I: achalasia with minimum esophageal pressurization, type II: achalasia with esophageal compression and type III: achalasia with spasm.

Previous studies have found that the pathological features of the esophageal muscular layers in participants with achalasia are degeneration of nerve plexus, reduction of interstitial cells of Cajal (ICCs) and infiltration of different inflammatory cells. Different subtypes of achalasia have different pathological characteristics and esophageal motility. Now, per-oral endoscopic myotomy (POEM) is a main therapy for participants with achalasia. Most studies have focused on the relationship between pathological features and motility characteristics of achalasia, but there are few studies on the relationship between pathological features and therapeutic effect of POEM.

This study will prospectively collect data of participants undergoing POEM for achalasia in Beijing Friendship Hospital, including demographic data, drug and surgical treatment data during hospitalization. All participants are required to obtain esophageal muscle biopsy for pathological examination during POEM. The participants will be followed up until 12 months for improvement in clinical symptoms.

DETAILED DESCRIPTION:
Achalasia is the most common motility disorder of esophagus, characterized by disorders of the lower esophageal sphincter (LES). Normal peristalsis of the esophagus is eliminated and replaced by synchronous or ineffective contraction. Based on high-resolution manometry (HRM), the participants with achalasia were categorized into 3 subtypes, type I: achalasia with minimum esophageal pressurization, type II: achalasia with esophageal compression and type III: achalasia with spasm.

Previous studies have found that the pathological features of the esophageal muscular layers in participants with achalasia are degeneration of nerve plexus, reduction of interstitial cells of Cajal (ICCs) and infiltration of different inflammatory cells. Different subtypes of achalasia have different clinical characteristics and esophageal motility. Studies have found that ganglion cells in type I participants are significantly reduced compared with type II participants, but the pattern is similar, which may indicate that type I achalasia represents the progression of type II achalasia. In addition, Achalasia is related to viral infection and autoimmune disease. Studies have shown that pathological biopsies of muscle in participants with achalasia show significantly increased rates of lymphocytes in tissues, as well as mast cells.

Now, per-oral endoscopic myotomy (POEM) is a main therapy for participants with achalasia. Most studies have focused on the relationship between pathological features and motility characteristics of achalasia, but there are few studies on the relationship between pathological features and therapeutic effect of POEM.

This study will prospectively collect data of participants undergoing POEM for achalasia in Beijing Friendship Hospital, including demographic data, drug and surgical treatment data during hospitalization. All participants are required to obtain esophageal muscle biopsy for pathological examination during POEM. The participants will be followed up until 12 months for improvement in clinical symptoms and gastroesophageal reflux after POEM.

ELIGIBILITY:
Inclusion Criteria:

* Participants with achalasia
* Age: 18 to 80 years
* Accept for the treatment of POEM
* Sign the informed consent

Exclusion Criteria:

* Participants under 18 years old
* Previously received treatment of achalasia, Barrett's esophagus, esophageal stricture, liver cirrhosis, and/or esophageal varices, tumors, allergic diseases and hiatal hernia.
* Use non-steroidal anti-inflammatory drugs, corticosteroids and other immunosuppressive agents.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with achalasia are hospitalized in Beijing Friendship Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-11 (Actual); Primary Completion 2024-04-16 (Estimated); Study Completion 2024-04-16 (Estimated)

PRIMARY OUTCOMES:
Eckardt score | 12months after POEM
  Eckardt score is used to assess the severity of symptoms in participants with achalasia. The Eckardt score evaluates weight loss, dysphagia, retrosternal pain, and reflux of achalasia. The maximum value is 12 and the minimum value is 0. Higher scores mean a worse outcome.

SECONDARY OUTCOMES:
GERDQ score | 12months after POEM
  GERDQ is a abbreviation of gastroesophageal reflux disease questionnaire. GERDQ score is used to assess the degree of gastroesophageal reflux after POEM. The maximum value is 18 and the minimum value is 0. Higher scores mean a worse outcome. Gastroesophageal reflux disease can be diagnosed if the GERDQ score is greater than or equal to 8.

CONTACTS AND LOCATIONS:
Overall Officials: Fandong Meng, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Investigators haven't decided which parts to share yet.

REFERENCES:
- [Background] Liu ZQ, Chen WF, Wang Y, Xu XY, Zeng YG, Lee Dillon D, Cheng J, Xu MD, Zhong YS, Zhang YQ, Yao LQ, Zhou PH, Li QL. Mast cell infiltration associated with loss of interstitial cells of Cajal and neuronal degeneration in achalasia. Neurogastroenterol Motil. 2019 May;31(5):e13565. doi: 10.1111/nmo.13565. Epub 2019 Mar 13. PMID 30868687

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05113173/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT05113173/ICF_001.pdf